CLINICAL TRIAL: NCT02150031
Title: Bacteraemia Secondary to Tooth Extraction: a Randomized Clinical Trial on Efficacy of Three Different Chlorhexidine Prophylaxis Protocols
Brief Title: Bacteraemia Secondary to Tooth Extraction: Chlorhexidine Prophylaxis Protocols
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, Inmaculada Tomas, Senior lecturer, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2008/202 CHX bacteraemia
Record Dates: First submitted 2014-05-16; First posted 2014-05-29 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Bacteremia; Tooth Extraction Status Nos
Keywords: prevention and control; chlorhexidine; therapeutic irrigation; mouthwashes; culture
MeSH Terms: conditions — Bacteremia | interventions — Chlorhexidine; Solutions; Lidocaine; Epinephrine; Anesthesia; Tooth Extraction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (Other): * Blood extraction using the intravenous access 18-22 gauge "angiocath" catheter (Becton Dickinson, Sparks, MD, USA) (at baseline, 30 seconds and 15 minutes after tooth extraction).
  * No prophylactic Chlorhexidine regimen.
  * Local anesthesia with lidocaine plus adrenaline (1:100,000).
  * Tooth extraction.
  Interventions: Procedure: Blood extraction; Drug: Lidocaine plus adrenaline; Procedure: Tooth extraction
- CHX-Mouthwash (Active Comparator): * Blood extraction using the intravenous access 18-22 gauge "angiocath" catheter (Becton Dickinson, Sparks, MD, USA)(at baseline, 30 seconds and 15 minutes after tooth extraction).
  * Mouthwash with 0.2% Chlorhexidine (10 ml for 1 minute) (Oraldine Perio®, Johnson and Johnson, Barcelona, Spain).
  * Local anesthesia with lidocaine plus adrenaline (1:100,000).
  * Tooth extraction.
  Interventions: Drug: 0.2% Chlorhexidine; Procedure: Blood extraction; Drug: Lidocaine plus adrenaline; Procedure: Tooth extraction
- CHX-MW/SUB_IR (Active Comparator): * Blood extraction using the intravenous access 18-22 gauge "angiocath" catheter (Becton Dickinson, Sparks, MD, USA) (at baseline, 30 seconds and 15 minutes after tooth extraction).
  * Mouthwash with 0.2% Chlorhexidine (10 ml for 1 minute) (Oraldine Perio®) and subgingival irrigation with 1% Chlorhexidine on the tooth to be extracted; the irrigation will be done with the Heraeus Citojet Intraligamental Syringe (Kulzer Heraeus S.A., Madrid, Spain) at six points on each tooth (3 points on the vestibular surface and 3 on the palatine surface).
  * Local anesthesia with lidocaine plus adrenaline (1:100,000).
  * Tooth extraction.
  Interventions: Drug: 0.2% Chlorhexidine; Drug: 1% Chlorhexidine; Procedure: Blood extraction; Drug: Lidocaine plus adrenaline; Procedure: Tooth extraction
- CHX-MW/SUPRA_IR (Active Comparator): * Blood extraction using the intravenous access 18-22 gauge "angiocath" catheter (Becton Dickinson, Sparks, MD, USA)(at baseline, 30 seconds and 15 minutes after tooth extraction).
  * Mouthwash with 0.2% Chlorhexidine (10 ml for 1 minute) (Oraldine Perio®) and then supragingival irrigation with 1% Chlorhexidine on the tooth to be extracted; the irrigation will be done continuously around the tooth to be extracted by a conventional syringe.
  * Local anesthesia with lidocaine plus adrenaline (1:100,000).
  * Tooth extraction.
  Interventions: Drug: 0.2% Chlorhexidine; Drug: 1% Chlorhexidine; Procedure: Blood extraction; Drug: Lidocaine plus adrenaline; Procedure: Tooth extraction

INTERVENTIONS:
Drug: 0.2% Chlorhexidine — mouthwash with 10 ml for 1 minute
  Other Names: OraldinePerio; Chlorhexidine 0.2%
  Arms: CHX-MW/SUB_IR; CHX-MW/SUPRA_IR; CHX-Mouthwash
Drug: 1% Chlorhexidine — subgingival irrigation
  Other Names: Normosept 1g/100ml sloution; Chlorhexidine 1%
  Arms: CHX-MW/SUB_IR
Drug: 1% Chlorhexidine — supragingival irrigation
  Other Names: Normosept 1g/100ml solution; Chlorhexidine 1%
  Arms: CHX-MW/SUPRA_IR
Procedure: Blood extraction — Blood extraction using an intravenous access at baseline, 30 seconds after antiseptic aplication, 30 seconds and 15 minutes after tooth extraction.
Drug: Lidocaine plus adrenaline — local anaesthesia using lidocaine plus adrenaline (1:100,000) no more than 2 cartridges.
  Other Names: anaesthesia
Procedure: Tooth extraction — dental extraction

SUMMARY:
The first time the American Heart Association (AHA) suggested that disinfection of the gingival sulcus be performed as a complement to antibiotic prophylaxis in patients considered to be at risk of Infective endocarditis (IE) was in their protocol for the prevention of IE published in 1977. This practice was included by the AHA and adopted by other expert committees such as the British Society for Antimicrobial Chemotherapy (BSAC) in subsequent prophylactic regimens. In 1992, the BSAC specified the presentation and concentration of chlorhexidine (CHX) that should be used before starting the dental procedure: 1% gel at the gingival margin or 0.2% mouthwash for five minutes. In 1997, the AHA recognised the need to use antiseptic mouthwashes (CHX or povidone iodine) prior to dental manipulations, although they recommended against the use of gingival irrigators and against the continuous use of antiseptics in order to avoid the selection of resistant micro-organisms In 2006, the BSAC recommended a single mouthwash with 0.2% CHX gluconate (10 ml for 1 minute) before performing dental procedures associated with bacteraemia in patients at risk of IE. In contrast, in 2007, the AHA recommended against the use of any antiseptic prophylaxis protocol.

In 2008, the National Institute for Health and Clinical Excellence of the United Kingdom recently performed a systematic review of the antimicrobial prophylaxis protocols for IE and reported that: "Oral chlorhexidine used as an oral rinse does not significantly reduce the level of bacteraemia following dental procedures". This conclusion was reached after analysis of numerous studies on the efficacy of prophylaxis with CHX for the prevention of post-dental manipulation bacteraemia. However, those studies presented significant methodological differences not only in the dental procedures performed, but also in the concentration of CHX applied and the method of application of the antiseptic solution (mouthwash and/or irrigation), making comparison of the results of the different series difficult.

There are few studies that have analysed the efficacy of the mouthwash of 0.2% CHX (the concentration recommended by the BSAC) in the prevention of post-extraction bacteraemia. Only one study analysed the combination of local irrigation and mouthwash with chlorhexidine before dental extraction, but with a really lower concentration of CHX, only 0.02%.

The objective of this study is to investigate the prevalence, duration and aetiology of bacteraemia secondary to a single tooth extraction after prophylaxis with different CHX protocols.

DETAILED DESCRIPTION:
The study group will be formed of patients undergoing tooth extraction under local anaesthesia in the Department of Stomatology and Maxillofacial Surgery of the Santo Antonio General Hospital (Oporto, Portugal).The following exclusion criteria will be applied: patients under 18 years of age; antibiotic treatment in the previous three months; routine use of oral antiseptics; and any type of congenital or acquired immunodeficiency or other disease that can favour the onset of infection or haemorrhagic complications. Applying these criteria and after a statistic power test, the sample will be 208 patients. The select patients will be attributed randomly a number of participation and they will be distributed into four groups:

* Control Group: 52 patients who will use no prophylactic chlorhexidine (CHX) regimen.
* CHX mouthwash group (CHX-MW group): 52 patients who will perform a mouthwash with 0.2% CHX (10 ml for 1 minute, BSAC recommendations) (Oraldine Perio®, Johnson and Johnson, Barcelona, Spain) before the tooth extraction.
* CHX mouthwash/subgingival irrigation group (CHX-MW/SUB_IR group): 52 patients who will perform a mouthwash with 0.2% CHX (10 ml for 1 minute) (Oraldine Perio®) and who then will undergo subgingival irrigation with 1% CHX on the tooth to be extracted; the irrigation will be done with the Heraeus Citojet Intraligamental Syringe (CIS) (Kulzer Heraeus S.A., Madrid, Spain) at six points on each tooth (3 points on the vestibular surface and 3 on the palatine surface).
* CHX mouthwash/supragingival irrigation group (CHX-MW/SUPRA_IR group): 52 patients who will perform a mouthwash with 0.2% CHX (10 ml for 1 minute) (Oraldine Perio®) and who then will undergo supragingival irrigation with 1% CHX on the tooth to be extracted; the irrigation will be done continuously around the tooth to be extracted by a conventional syringe.

The mouthwash and subgingival or supragingival irrigation will be performed before injection of the local anaesthetic.

After recording the sex and age of each patient, a single dentist will perform an intraoral examination 2 days before the intervention, collecting the following information: plaque deposits (simplified Greene and Vermillion oral hygiene index) , calculus deposits (Ramfjord calculus index), presence of gingival bleeding (Löe and Silness gingival index), depth of periodontal pockets (Ramfjord index), degree of tooth mobility (Ramfjord tooth mobility index), number of caries (including root remnants), and presence of submucosal abscesses, fistulae and periapical foci detected clinically and/or radiologically. Each patient will be assigned an overall oral health status using a scale designed by the authors and published previously; the scale incorporates dental and periodontal health criteria.

Local anaesthesia will be administered to all patients using conventional techniques (regional block and/or infiltration). The anaesthetic will be lidocaine plus adrenaline (1:100,000) and not more than 2 cartridges in any patient.

The prevalence of baseline bacteraemia will be determined by collection of a peripheral venous blood sample (10 ml) from each patient before performing any manipulation. The prevalence of bacteraemia secondary to a mouthwash and subgingival or supragingival irrigation will be determined by the collection of a peripheral blood sample (10 ml) 30 seconds after each of these actions. Further samples (10 ml) will be drawn 30 seconds and 15 minutes after completion of the tooth extraction in order to determine the prevalence and duration of post-extraction bacteraemia.

Intravenous access will established using an 18-22 gauge "angiocath" catheter (Becton Dickinson, Sparks, MD, USA) inserted in the antecubital fossa or dorsum of the hand after disinfection of the area with alcohol and povidone iodine. The catheter will be flushed with 3 ml of saline after each extraction and the first 2 ml of blood was discarded. Equal volumes of each sample will be inoculated into two bottles containing aerobic and anaerobic culture media (Bactec Plus, Becton Dickinson), and the bottles will be immediately transferred to the laboratory. The whole process of manipulation and transport of the samples will be performed in accordance with the recommendations of the Spanish Society of Infectious Diseases and Clinical Microbiology.

The blood culture bottles into which the blood samples will be injected and processed in the Bactec 9240 (Becton Dickinson). Gram stain will be performed on all positive cultures. The positive aerobic blood cultures will be subcultured on blood agar and chocolate agar in an atmosphere with 5%-10% CO2, and on MacConkey agar under aerobic conditions. The same protocol will be used for the positive anaerobic blood cultures but include subculture on Schaedler agar and incubation under anaerobic conditions. The bacteria isolated will be identified using the battery of biochemical tests provided by the Vitek system (bioMérieux Inc., Hazelwood, Missouri, USA) for gram-positive bacteria, Neisseria spp./Haemophilus spp. and obligate anaerobic bacteria. Applying the Ruoff criteria, Streptococcus viridans will be classified into five groups: mutans, salivarius, bovis, anginosus and mitis.

ELIGIBILITY:
Inclusion Criteria:

* with need for dental extraction

Exclusion Criteria:

* patients under 18 years of age
* antibiotic treatment in the previous three months
* routine use of oral antiseptics
* any type of congenital or acquired immunodeficiency or other disease that could favour the onset of infection or haemorrhagic complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2010-12; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Changes in the prevalence of bacteraemia | before and 30 seconds after the antiseptic aplication and 30 seconds and 15 minutes after dental extraction.
  Presence of bacteria and how long it lasts in the blood stream.

CONTACTS AND LOCATIONS:
Overall Officials: Inmaculada Tomas, Principal Investigator — Senior lecturer at University of Santiago de Compostela
Locations (2):
- Department of Stomatology and Maxillofacial Surgery of the Santo Antonio General Hospital, Porto, Porto District, Portugal
- Department of Stomatology University of Santiago de Compostela, Santiago de Compostela, Galicia/A Coruña, Spain

REFERENCES:
- [Background] Tomas I, Alvarez M, Limeres J, Tomas M, Medina J, Otero JL, Diz P. Effect of a chlorhexidine mouthwash on the risk of postextraction bacteremia. Infect Control Hosp Epidemiol. 2007 May;28(5):577-82. doi: 10.1086/516663. Epub 2007 Apr 5. PMID 17464918
- [Background] Tomas I, Alvarez M, Limeres J, Potel C, Medina J, Diz P. Prevalence, duration and aetiology of bacteraemia following dental extractions. Oral Dis. 2007 Jan;13(1):56-62. doi: 10.1111/j.1601-0825.2006.01247.x. PMID 17241431
- [Background] Benitez-Paez A, Alvarez M, Belda-Ferre P, Rubido S, Mira A, Tomas I. Detection of transient bacteraemia following dental extractions by 16S rDNA pyrosequencing: a pilot study. PLoS One. 2013;8(3):e57782. doi: 10.1371/journal.pone.0057782. Epub 2013 Mar 4. PMID 23469240
- [Background] Pineiro A, Tomas I, Blanco J, Alvarez M, Seoane J, Diz P. Bacteraemia following dental implants' placement. Clin Oral Implants Res. 2010 Sep;21(9):913-8. doi: 10.1111/j.1600-0501.2010.01928.x. PMID 20701619
- [Derived] Barbosa M, Prada-Lopez I, Alvarez M, Amaral B, de los Angeles CD, Tomas I. Post-tooth extraction bacteraemia: a randomized clinical trial on the efficacy of chlorhexidine prophylaxis. PLoS One. 2015 May 8;10(5):e0124249. doi: 10.1371/journal.pone.0124249. eCollection 2015. PMID 25955349